CLINICAL TRIAL: NCT01780298
Title: A Biomarker Study to Compare Gene and Protein Expression Profiles in Four Separate Groups of Subjects Including COPD Cases (GOLD Stage 1-2 and Current Smokers With a ≥ 10 Pack Year Smoking History) and Three Control Groups of Matched Non-smoking Subjects (Never Smoked), Ex-smokers and Current Smokers, to Identify Novel Biomarkers, to Assess Standard Biomarkers of Inflammation and to Compare Inflammatory Cell Responses and Selected Markers of Inflammation in Blood, Induced Sputum and Nasal Samples.
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Biomarker Identification Study
Status: Completed | Type: Observational
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: QASMC 202
Record Dates: First submitted 2013-01-21; First posted 2013-01-31 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: COPD
Keywords: COPD; Biomarkers; Cigarette Smoke; Lung Inflammation; FEV; Sputum
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cigarette Smoking; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Proteomic investigations: Induced Sputum
  Transcriptomics investigations (mRNA and micro RNA): Whole Blood, Nasal Scrapes, Induced sputum cell pellet
  Genomic DNA sequencing: Whole blood
  Lipidomics: Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: COPD GOLD Stage 1-2: Subjects with a clinical diagnosis of COPD, according to the GOLD guidelines (Stages 1-2), who are current smokers with at least a 10 pack-year smoking history.
- Group 2: Current Cigarette Smokers: Subjects who are current smokers with at least a 10 pack-year smoking history, and matched to the COPD cases by ethnicity, gender and age (within 5 years).
- Group 3: Ex-Smokers: Subjects who are ex-smokers with at least a 10 pack-year smoking history who have not smoked for at least one year, and matched to the COPD cases by ethnicity, gender and age (within 5 years).
- Group 4: Never Smokers: Subjects who have never smoked (non-smokers), and matched to the COPD cases by ethnicity, gender and age (within 5 years).

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a common inflammatory disease of the airway affecting approximately 10% of individuals aged 40 years or more with a smoking history. The disease is characterized by an increase in numbers of airway white blood cells (neutrophils, lymphocytes and monocytes). Stimulation of white blood cells results in the release of different agents of inflammation. Some of these agents give an indication of the presence or severity of a disease when measured.

This case control study will be conducted at The Heart Lung Centre, London, UK. The study aims to determine biomarkers for the differentiation of subjects with COPD (GOLD Stage 1-2 and who are current smokers with a ≥ 10 pack year smoking history) and three matched control groups: one of non-smoking subjects (never smoked), one of ex-smokers and one of current smokers. COPD subjects will be matched to the non-COPD subjects by gender, age and ethnicity.

The study will include a range of physiological measurements including lung function, computerized tomography scans (CT scans), cardio pulmonary exercise test and computerized multichannel lung sounds analysis (Stethographics). In addition, lung inflammation will be assessed by cellular and molecular biomarkers using e.g. transcriptomics and proteomics technologies.

DETAILED DESCRIPTION:
At the screening visit, subject consent will be obtained prior to conducting any study related procedures. Informed consent may be obtained on registration/review visit at the Centre where it is conducted and thus prior to visit 1.

The screening visit will involve obtaining demographic data and medical history information as well as performing safety assessments such as vital sign measurements, electrocardiogram (ECG), and clinical laboratory tests. An induced sputum sample will be obtained to ensure that subjects can produce an adequate sputum sample. Smokers will receive information on smoking cessation at the screening visit and follow-up telephone call.

Subjects will come back to the center on up to four further occasions if they meet the inclusion/exclusion criteria at screening:

* visit 2: 4 to 21 days after screening,
* visit 3: 3-14 days post visit 2, and
* visit 4: 3-14 days post visit 3.

A follow-up telephone call will be conducted 3-10 days post visit 4.

ELIGIBILITY:
Inclusion Criteria

* Provision of signed written informed consent which includes genetic consent.
* Ability to comply with study procedures.
* Males and females aged 40-70 years inclusive.
* Have a body mass index (BMI) between 18 and 35 kg/m2 inclusive and minimum body weights of 50 kg.
* Have a normal physical examination, and have normal laboratory values, 12-lead ECG and vital signs (blood pressure, heart rate and respiratory rate), unless the Investigator considers an abnormality as not clinically significant.
* Ability to perform reproducible spirometry according to the American Thoracic Society and the European Respiratory Society (ATS/ERS) guidelines (American Thoracic Society, 2005).
* Ability to produce a minimum 0.1 gram sputum sample after induction with inhaled hypertonic saline.

Additional Inclusion Criteria COPD Group

* A clinical diagnosis of COPD according to the GOLD guidelines (stage 1-2).
* Current smokers with ≥10 pack-year smoking history.
* Demonstrate a post-bronchodilator ratio between forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) of <70 % and FEV1 ≥50 % of predicted normal.

Additional Inclusion Criteria Non-Smokers Group

* Have never smoked tobacco products.
* Demonstrate normal lung function by post bronchodilator FEV1 ≥80 % of predicted normal, with no evidence of airway obstruction FEV1/FVC ratio ≥70 %.
* Have a sputum eosinophilia <2 % and a sputum neutrophilia <80 % from the sample collected at visit 1 (Belda et al., 2000).

Additional Inclusion Criteria Smokers Group

* Be current smokers with defined smoking history of ≥10 pack years.
* Have normal lung function by post bronchodilator FEV1 ≥80 % of predicted normal, with no evidence of airway obstruction FEV1/FVC ratio ≥70 %.

Additional Inclusion Criteria Ex-Smokers Group

* Be ex-smokers, with defined smoking history of ≥10 pack years and to have quit smoking at least 1 year before entering the study.
* Have normal lung function by post bronchodilator FEV1 ≥80 % of predicted normal, with no evidence of airway obstruction FEV1/FVC ratio ≥70 %.

Exclusion Criteria:

* Current evidence or recent history of any clinically significant disease or abnormality (other than COPD in the subjects with COPD group), which in the opinion of the Investigator, would put the subject at risk, or which would compromise the quality of the study data, including but not limited, to cardiovascular disease, myocardial infarction, cardiac failure, uncontrolled hypertension, life-threatening arrhythmias, uncontrolled diabetes, neurologic or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities.
* Females with a positive pregnancy test at visit 1 or 3.
* Females currently breastfeeding.
* Involvement in the planning and conduct of the study.
* Surgery or significant trauma within 3 months of visit 1.
* History of tuberculosis or other non-specific pulmonary diseases such as asthma.
* Symptoms, signs or laboratory findings suggestive of an ongoing infective illness as judged by the Investigator at visit 1 or 2.
* Participation in any clinical study with an investigational drug in the 4 months prior to visit 1, or participation in a study with a new formulation of a marketed drug in the 3 months prior to visit 1, or participation in a methodology study in the month prior to visit 1.
* Symptoms of any clinically significant illness within 2 weeks prior to visit 1.
* A significant history of alcohol abuse or consumption of more than the recommended units of alcohol per week (28 units for males and 21 units for females).
* A significant history of drug abuse (including benzodiazepines) or a positive test of drug abuse test at visit 1.
* Subjects, who in the opinion of the Investigator should not, for safety or compliance reasons, participate in the study.
* Use of prohibited medications.
* Subjects who have a first degree relative (parents, sibling or child) already enrolled in the study.

Additional Exclusion Criteria - subjects with COPD

* Recent history of hospitalization due to an exacerbation of airway disease within 3 months of the screening visit or subjects with need for increased treatments for COPD within 6 weeks prior to the screening visit.
* Prior lung volume reduction surgery or history of chest/lung irradiation.
* Regular use of daily oxygen therapy.
* Long standing history and primary diagnosis of asthma.
* Use of systemic steroids within 3 months prior to the screening visit.
* Respiratory tract infection within 6 weeks prior to the screening visit.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, male and female subjects aged between 40-70 years will be included. All subjects must be matched by ethnicity, gender and age (within 5 years) of the subjects with COPD recruited in the study.
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leaker, MD, Principal Investigator — Heart Lung Centre, Queen Anne Street Medical Centre
Locations (1):
- Heart Lung Centre, Queen Anne Street Medical Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data for transcriptomics (sputum and nasal scrapes) and proteomics (sputum) are published and available via the following links:
  * Sputum transcriptomics:
  http://www.ebi.ac.uk/arrayexpress/experiments/E-MTAB-3604/
  * Sputum proteomics:
  http://www.ebi.ac.uk/pride/archive/projects/PXD001977
  * Nasal scrapes transcriptomics:
  http://www.ebi.ac.uk/arrayexpress/experiments/E-MTAB-4015/
  * Blood transcriptomics:
  The link to the Array Express database will be provided upon online publication
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.
URL: https://doi.org/10.12688/f1000research.11698.2

REFERENCES:
- [Result] Titz B, Sewer A, Schneider T, Elamin A, Martin F, Dijon S, Luettich K, Guedj E, Vuillaume G, Ivanov NV, Peck MJ, Chaudhary NI, Hoeng J, Peitsch MC. Alterations in the sputum proteome and transcriptome in smokers and early-stage COPD subjects. J Proteomics. 2015 Oct 14;128:306-20. doi: 10.1016/j.jprot.2015.08.009. Epub 2015 Aug 22. PMID 26306861
- [Result] Martin F, Talikka M, Hoeng J, Peitsch MC. Identification of gene expression signature for cigarette smoke exposure response--from man to mouse. Hum Exp Toxicol. 2015 Dec;34(12):1200-11. doi: 10.1177/0960327115600364. PMID 26614807
- [Result] Chaudhary N, Luettich K, Peck MJ, Pierri E, Felber-Medlin L, Vuillaume G, Leroy P, Hoeng J, Peitsch MC. Physiological and biological characterization of smokers with and without COPD. F1000Res. 2017 Jun 13;6:877. doi: 10.12688/f1000research.11698.2. eCollection 2017. PMID 29862011
- [Derived] Titz B, Luettich K, Leroy P, Boue S, Vuillaume G, Vihervaara T, Ekroos K, Martin F, Peitsch MC, Hoeng J. Alterations in Serum Polyunsaturated Fatty Acids and Eicosanoids in Patients with Mild to Moderate Chronic Obstructive Pulmonary Disease (COPD). Int J Mol Sci. 2016 Sep 20;17(9):1583. doi: 10.3390/ijms17091583. PMID 27657052
- See also: Sputum transcriptomics — http://www.ebi.ac.uk/arrayexpress/experiments/E-MTAB-3604/
- See also: Sputum proteomics — http://www.ebi.ac.uk/pride/archive/projects/PXD001977
- See also: Nasal scrapes transcriptomics — http://www.ebi.ac.uk/arrayexpress/experiments/E-MTAB-4015/
- Available data/document: Individual Participant Data Set — https://doi.org/10.12688/f1000research.11698.2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject enrolled): 01 July 2011
Period: Overall Study
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Started | 62 | 65 | 64 | 61
Completed | 60 | 60 | 60 | 60
Not Completed | 2 | 5 | 4 | 1
Not completed — Physician Decision | 1 | 5 | 1 | 1
Not completed — Subject not matched | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers | Total
Number analyzed (Participants) | 62 | 65 | 64 | 61 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.161 (7.159) | 55.308 (6.908) | 56.344 (7.392) | 55.459 (7.453) | 56.063 (7.223)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 27 | 26 | 107
  Male | 37 | 36 | 37 | 35 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 4
  White | 60 | 64 | 63 | 60 | 247
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.461 (3.700) | 27.568 (3.657) | 27.333 (3.558) | 26.479 (3.719) | 26.972 (3.670)
Number of Cigarettes Smoked Per Day [Mean (Standard Deviation); unit: Cig/day] | 20.611 (9.412) | 17.319 (7.541) | 22.422 (9.135) | 0 (0) | 15.233 (11.611)
Pack-year [Mean (Standard Deviation); unit: Pack-year] | 44.770 (22.019) | 33.404 (14.577) | 28.535 (13.330) | 0 (0) | 26.878 (21.977)
Weekly Consumption of Alcohol [Mean (Standard Deviation); unit: Units of alcohol] — The weekly consumption of alcohol is expressed in "Units of alcohol".
  Units of alcohol are used as a measure to quantify the actual alcoholic content within a given volume of an alcoholic beverage, in order to provide guidance on total alcohol consumption. One unit of alcohol is defined as 10 milliliters (8 grams) of pure alcohol.
  At the time this study was planned and conducted, the recommended units of alcohol not to be exceeded per week were 28 units for males and 21 units for females.
  Units of alcohol | 6.694 (7.662) | 5.923 (6.310) | 8.445 (7.097) | 5.775 (6.711) | 6.717 (6.998)

OUTCOME MEASURES:

1. Primary Outcome: Spirometry Measurement: Percentage of Predicted Forced Expiratory Volume in 1 Second (FEV1 %Pred)
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: percent of predicted FEV1
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
percent of predicted FEV1 | 75.572 [70.905 to 80.239] | 100.837 [97.801 to 103.873] | 108.311 [105.102 to 111.519] | 111.849 [108.258 to 115.440]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Pairwise comparisons obtained by 2-sided paired t-test (COPD subjects are paired to the non-COPD subjects by gender, age and ethnicity); Mean Difference (Final Values) = -36.278, 95% CI 2-sided [-42.203 to -30.352] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -32.739, 95% CI 2-sided [-38.418 to -27.060] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -25.265, 95% CI 2-sided [-31.081 to -19.449] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.1504, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.538, 95% CI 2-sided [-8.398 to 1.321] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.0002, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.474, 95% CI 2-sided [-11.207 to -3.741] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.013, 95% CI 2-sided [-15.979 to -6.046] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

2. Primary Outcome: Gas Transfer: Percentage of Predicted Total Diffusing Capacity of the Lungs for Carbon Monoxide (TLCO %Pred)
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: percent predicted TLCO
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
percent predicted TLCO | 66.158 [61.981 to 70.334] | 80.264 [77.043 to 83.485] | 90.710 [87.134 to 94.286] | 93.768 [90.664 to 96.873]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -27.611, 95% CI 2-sided [-32.249 to -22.973] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -24.553, 95% CI 2-sided [-29.501 to -19.604] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.107, 95% CI 2-sided [-19.043 to -9.170] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0983, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.058, 95% CI 2-sided [-6.702 to 0.585] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.446, 95% CI 2-sided [-13.845 to -7.047] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.504, 95% CI 2-sided [-17.302 to -9.707] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

3. Primary Outcome: Impulse Oscillometry (IOS) Measurements: Percentage of Predicted Central Airway Resistance at 5Hz (R5 %Pred)
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: percent predicted R5
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
percent predicted R5 | 130.118 [119.600 to 140.637] | 109.458 [102.529 to 116.386] | 103.581 [97.437 to 109.724] | 89.671 [83.477 to 95.865]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 40.448, 95% CI 2-sided [28.374 to 52.521] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 26.538, 95% CI 2-sided [14.890 to 38.185] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p = 0.0018, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 20.661, 95% CI 2-sided [7.997 to 33.324] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0015, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 13.910, 95% CI 2-sided [5.534 to 22.286] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.1847, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.877, 95% CI 2-sided [-2.886 to 14.639] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 19.787, 95% CI 2-sided [9.536 to 30.038] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

4. Primary Outcome: Impulse Oscillometry (IOS) Measurements: Percentage of Predicted Reactance at 5 Hz (X5 % Pred)
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: percent predicted X5
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
percent predicted X5 | 2808.259 [-794.944 to 6411.462] | 411.670 [-139.923 to 963.263] | 491.128 [41.793 to 940.464] | 5787.984 [-902.669 to 12478.637]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.1981, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2979.725, 95% CI 2-sided [-7560.258 to 1600.808] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.1956, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2317.131, 95% CI 2-sided [-1224.786 to 5859.048] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p = 0.2077, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2396.589, 95% CI 2-sided [-1367.692 to 6160.870] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.1154, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5296.856, 95% CI 2-sided [-11930.190 to 1336.478] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.8095, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -79.458, 95% CI 2-sided [-736.151 to 577.234] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.1113, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5376.314, 95% CI 2-sided [-12030.714 to 1278.085] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

5. Primary Outcome: Impulse Oscillometry (IOS) Measurements: Resonant Frequency (Fres)
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: Hz
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
Hz | 17.816 [16.588 to 19.043] | 14.362 [13.513 to 15.210] | 12.971 [12.083 to 13.859] | 11.800 [10.942 to 12.659]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.015, 95% CI 2-sided [4.510 to 7.521] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.845, 95% CI 2-sided [3.379 to 6.310] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.454, 95% CI 2-sided [1.923 to 4.984] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0418, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.171, 95% CI 2-sided [0.045 to 2.296] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.0357, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.391, 95% CI 2-sided [0.096 to 2.686] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.562, 95% CI 2-sided [1.303 to 3.820] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

6. Primary Outcome: Stethographics Measurements: Non-Weighted Acoustic Chronic Obstructive Pulmonary Disease Scores (ACOPDS)
Description: Stethographics analysis was performed using the 16-channel lung sound analyzer system STG1602 (Stethographics, Boston, MA, USA) following the supplier's recommendations.
  Lung sound data are obtained from an intermediate deeper-than-normal breath (pattern 2; P2). Each breath pattern is recorded for a minimum of 30 seconds allowing 3 to 6 breaths to be taken, with measurements completed over 3 to 4 minutes.
  Each of the 16 parameters derived from one measurement are evaluated and a score from 0 to 10 is assigned based on the value of the individual parameter. The total standard Acoustic COPD Score (ACOPDS) is calculated as the sum of the individual score for each parameter, which permits a maximum score of 160.
  Although this stethographics analysis system was considered experimental, a higher score was associated with poor health outcomes and a lower score with a better health state.
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
score on a scale | 47.983 [42.723 to 53.244] | 18.817 [14.467 to 23.166] | 12.192 [9.025 to 15.358] | 8.350 [6.187 to 10.513]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 39.633, 95% CI 2-sided [33.964 to 45.302] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 35.792, 95% CI 2-sided [29.761 to 41.822] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 29.167, 95% CI 2-sided [23.445 to 34.888] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0418, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.842, 95% CI 2-sided [0.147 to 7.536] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.0084, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6.625, 95% CI 2-sided [1.763 to 11.487] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.467, 95% CI 2-sided [5.888 to 15.045] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

7. Primary Outcome: Dyspnoea Assessment: Modified Medical Research Council (MMRC) Dyspnoea Scale
Description: The MMRC scale uses a simple grading system to assess a subject's level of dyspnea (shortness of breath).
  Subjects were asked to grade the degree of breathlessness related to activities by choosing 1 of the following answers:
  * 0: Not troubles by breathlessness except on strenuous exercise
  * 1: Short of breath when hurrying or walking up a slight hill
  * 2: Walks slower than contemporaries on the level because of breathlessness, or has to stop for breath when walking at own pace
  * 3: Stops for breath after about 100 meters or after a few minutes on the level
  * 4: Too breathless to leave the house, or breathless when dressing or undressing.
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 completed the study, but 235 were included in the analysis population as data were missing for 5 subjects:
  * 3 subjects in the group "COPD GOLD stage 1-2"
  * 1 subject in the group "Ex-smokers"
  * 1 subject in the group "Never smokers"
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 57 | 60 | 59 | 59
units on a scale | 1.053 [0.821 to 1.285] | 0.417 [0.272 to 0.562] | 0.186 [0.073 to 0.300] | 0.119 [-0.001 to 0.238]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.929, 95% CI 2-sided [0.654 to 1.203] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.875, 95% CI 2-sided [0.609 to 1.141] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.649, 95% CI 2-sided [0.386 to 0.912] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.3985, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.069, 95% CI 2-sided [-0.093 to 0.231] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.0267, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.220, 95% CI 2-sided [0.026 to 0.414] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0036, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.305, 95% CI 2-sided [0.104 to 0.506] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

8. Primary Outcome: Prediction of Mortality and Hospitalizations: Modified BODE Index (mBODE)
Description: The BODE Index is a 10-point scale to assess prognostic factors in COPD patients. Body mass index ("B"), airway obstruction ("O"), dyspnea ("D"), and exercise tolerance ("E") are each graded on a 4 point scale (0 to 3), except body mass index (0 or 1) . The final BODE Index value is the sum of the scores for each prognostic factor, where a higher BODE score indicates a higher risk of death.
  The modified BODE (mBODE) index as defined by Lopez-Campos (2010) was used in this study, and is composed of the following factors:
  * Body mass index: (0 or 1)
  * Degree of airflow obstruction (FEV1% Pred): (0 to 3)
  * Functional dyspnea (MMRC Dyspnoea Scale): (0 to 3)
  * Exercise capacity (VO2max): (0 to 3)
  Lopez-Campos, José Luis, et al. "Modified BODE indexes: Agreement between multidimensional prognostic systems based on oxygen uptake." International Journal of Chronic Obstructive Pulmonary Disease (2010): 133-140.
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 completed the study, but 233 were included in the analysis population as data were missing for 7 subjects:
  * 4 subjects in the group "COPD GOLD stage 1-2"
  * 1 subject in the group "Current cigarette smokers"
  * 1 subject in the group "Ex-smokers"
  * 1 subject in the group "Never smokers"
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 56 | 59 | 59 | 59
score on a scale | 2.357 [1.998 to 2.716] | 1.254 [1.035 to 1.474] | 1.051 [0.827 to 1.275] | 0.763 [0.555 to 0.970]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.564, 95% CI 2-sided [1.179 to 1.949] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.291, 95% CI 2-sided [0.924 to 1.658] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.073, 95% CI 2-sided [0.724 to 1.421] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0282, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.276, 95% CI 2-sided [0.031 to 0.521] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.1223, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.207, 95% CI 2-sided [-0.057 to 0.471] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.492, 95% CI 2-sided [0.273 to 0.710] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

9. Primary Outcome: High-Resolution Computerised Tomography (HRCT) of the Chest
Description: CT scans were assessed by two radiologists. A scoring system from 0 to 4 was applied, depending upon the component:
  1. Extent of disease (emphysema): 0=absent, 1=mild, 2=moderate, 3=severe, 4=very severe
  2. Severity of bronchial dilatation: 0=none; 1=mild (1.5x to 2.5x diameter of pulmonary artery); 2=severe (>2.5x diameter of pulmonary artery)
  3. Traction bronchiectasis: 0=none; 1=mild (1.5x to 2.5x diameter); 2=severe (>2.5x diameter).
  4. Total bronchiectasis score derived by adding the bronchial dilatation and traction bronchiectasis scores
  5. Bronchial wall thickening: 0=none; 1=0.5x; 2=0.5-1x; 3= >1x the diameter of the adjacent pulmonary artery
  6. Small airways disease: 0=absent, 1=mild, 2=moderate, 3=severe and 4=very severe
  The total score (higher score indicated a poor outcome) was derived from the mean of all scores. This is described in Chaudhary, Nveed, et al. "Physiological and biological characterization of smokers with and without COPD." F1000Research 6 (2017).
Time Frame: Up to 59 days
Population: Of the 252 enrolled subjects, 240 (60 per group) completed the study, and were included in the analysis population.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Number analyzed (Participants) | 60 | 60 | 60 | 60
score on a scale | 0.939 [0.867 to 1.011] | 0.803 [0.723 to 0.884] | 0.683 [0.613 to 0.753] | 0.567 [0.488 to 0.646]
Statistical Analysis 1: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.372, 95% CI 2-sided [0.269 to 0.478] — Difference Group 1 (COPD) - Group 4 (Never smokers)
Statistical Analysis 2: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 3: Ex-Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.256, 95% CI 2-sided [0.158 to 0.354] — Difference Group 1 (COPD) - Group 3 (Ex-smokers)
Statistical Analysis 3: Comparison: Group 1: COPD GOLD Stage 1-2 vs Group 2: Current Cigarette Smokers; Test type: Superiority or Other; p = 0.0199, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.136, 95% CI 2-sided [0.022 to 0.249] — Difference Group 1 (COPD) - Group 2 (Current cigarette smokers)
Statistical Analysis 4: Comparison: Group 3: Ex-Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p = 0.0247, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.117, 95% CI 2-sided [0.015 to 0.218] — Difference Group 3 (Ex-smokers) - Group 4 (Never smokers)
Statistical Analysis 5: Comparison: Group 2: Current Cigarette Smokers vs Group 3: Ex-Smokers; Test type: Superiority or Other; p = 0.0204, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.120, 95% CI 2-sided [0.019 to 0.221] — Difference Group 2 (Current cigarette smokers) - Group 3 (Ex-smokers)
Statistical Analysis 6: Comparison: Group 2: Current Cigarette Smokers vs Group 4: Never Smokers; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.237, 95% CI 2-sided [0.127 to 0.347] — Difference Group 2 (Current cigarette smokers) - Group 4 (Never smokers)

10. Other Pre Specified Outcome: Total Leukocytes and Differential Leukocytes Count in Sputum
Description: Results are available at:
  Titz B, Sewer A, Schneider T, Elamin A, Martin F, Dijon S, Luettich K, Guedj E, Vuillaume G, Ivanov NV, Peck MJ, Chaudhary NI, Hoeng J, Peitsch MC.
  Alterations in the sputum proteome and transcriptome in smokers and early-stage COPD subjects. J Proteomics. 2015 Oct 14;128:306-20. doi: 10.1016/j.jprot.2015.08.009. Epub 2015 Aug 22.
  PMID: 26306861
Time Frame: Up to 59 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Protein Markers as Determined by Proteomics Analysis of Induced Sputum
Description: as for outcome 10
Time Frame: Up to 59 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Lipid Markers as Determined by Lipidomic Analysis of Blood Samples
Description: Reference to be provided upon publication.
Time Frame: Up to 59 days
Reporting Status: Not Posted

13. Other Pre Specified Outcome: mRNA and miRNA (Transcriptomics) Derived From Induced Sputum
Description: as for outcome 10
Time Frame: Up to 59 days
Reporting Status: Not Posted

14. Other Pre Specified Outcome: mRNA and miRNA (Transcriptomics) Derived From Leukocytes Obtained From Blood Samples
Description: Results are available at:
  Martin F, Talikka M, Hoeng J, Peitsch MC. Identification of gene expression signature for cigarette smoke exposure response--from man to mouse. Hum Exp Toxicol. 2015 Dec;34(12):1200-11. doi: 10.1177/0960327115600364
  PMID: 26614807
Time Frame: Up to 59 days
Reporting Status: Not Posted

15. Other Pre Specified Outcome: mRNA and miRNA (Transcriptomics) Derived From Nasal Epithelial Cells Obtained by Nasal Scrapes
Description: Reference to be provided upon publication.
Time Frame: Up to 59 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the informed consent form until the end of the study.
Description: The safety analysis was performed on the Study Population. As there was no investigational product, this was defined as all subjects who were enrolled into the study
Arm/Group | Group 1: COPD GOLD Stage 1-2 | Group 2: Current Cigarette Smokers | Group 3: Ex-Smokers | Group 4: Never Smokers
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/65 | 0/64 | 0/61
Other Adverse Events (participants affected / at risk) | 42/62 | 51/65 | 35/64 | 40/61
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: COPD GOLD Stage 1-2 (N=62) | Group 2: Current Cigarette Smokers (N=65) | Group 3: Ex-Smokers (N=64) | Group 4: Never Smokers (N=61)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 5 (5)
Computerised tomogram abnormal (Investigations) | 12 (12) | 28 (28) | 15 (15) | 24 (24)
Liver scan abnormal (Investigations) | 6 (6) | 0 (0) | 1 (1) | 2 (2)
Pulmonary function challenge test abnormal (Investigations) | 9 (9) | 16 (16) | 12 (12) | 15 (15)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 12 (12) | 7 (7) | 4 (4)
Headache (Nervous system disorders) | 10 (10) | 6 (6) | 4 (4) | 7 (7)
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.